CLINICAL TRIAL: NCT00184210
Title: HR MAS MR Spectroscopy of Breast Cancer Tissue
Brief Title: Magnetic Resonance (MR) Spectroscopy of Breast Cancer Tissue
Status: Terminated | Type: Observational
Why Stopped: the actual primary goal - establishment of an approved tissue biobank - was reached. 1000 tissue samples were collected. No motivation at this time for continuation as originally planned
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: The Research Council of Norway (Other); The Norwegian Women´s Public Health Association (Other)
Responsible Party: Sponsor
Other Study IDs: 154080/I30
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Breast Neoplasms
Keywords: Magnetic Resonance Spectroscopy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer tissue is collected from women undergoing scheduled surgery for breast cancer. The tissue specimen are analyzed by MR spectroscopy. After MR, the intact tissue specimen can be analyzed by other methods, such as histopathology.

The MR spectral profiles are compared to clinical findings such as the patients diagnosis, lymph node status and tumor size.

ELIGIBILITY:
Inclusion Criteria:

* Palpable breast cancer lesion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women in surgery for breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2000-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
MRimage of breast cancer tissue | 0 hour

CONTACTS AND LOCATIONS:
Overall Officials: Tone F Bathen, PhD, Study Chair — Norwegian University of Technology and Science
Locations (1):
- Norwegian University of Technology and Science, Trondheim, Norway

REFERENCES:
- [Result] Sitter B, Sonnewald U, Spraul M, Fjosne HE, Gribbestad IS. High-resolution magic angle spinning MRS of breast cancer tissue. NMR Biomed. 2002 Aug;15(5):327-37. doi: 10.1002/nbm.775. PMID 12203224
- [Result] Sitter B, Lundgren S, Bathen TF, Halgunset J, Fjosne HE, Gribbestad IS. Comparison of HR MAS MR spectroscopic profiles of breast cancer tissue with clinical parameters. NMR Biomed. 2006 Feb;19(1):30-40. doi: 10.1002/nbm.992. PMID 16229059
- [Result] Bathen TF, Jensen LR, Sitter B, Fjosne HE, Halgunset J, Axelson DE, Gribbestad IS, Lundgren S. MR-determined metabolic phenotype of breast cancer in prediction of lymphatic spread, grade, and hormone status. Breast Cancer Res Treat. 2007 Aug;104(2):181-9. doi: 10.1007/s10549-006-9400-z. Epub 2006 Oct 24. PMID 17061040
- [Result] Sitter B, Bathen TF, Singstad TE, Fjosne HE, Lundgren S, Halgunset J, Gribbestad IS. Quantification of metabolites in breast cancer patients with different clinical prognosis using HR MAS MR spectroscopy. NMR Biomed. 2010 May;23(4):424-31. doi: 10.1002/nbm.1478. Epub 2010 Jan 25. PMID 20101607
- [Result] Giskeodegard GF, Grinde MT, Sitter B, Axelson DE, Lundgren S, Fjosne HE, Dahl S, Gribbestad IS, Bathen TF. Multivariate modeling and prediction of breast cancer prognostic factors using MR metabolomics. J Proteome Res. 2010 Feb 5;9(2):972-9. doi: 10.1021/pr9008783. PMID 19994911